CLINICAL TRIAL: NCT03127410
Title: Predictive Validity of Lumbopelvic Stress Tests to Determine Those Who Will Benefit From Lumbar Traction: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Woman's University (Other)
Responsible Party: Principal Investigator, Kelli Brizzolara, Assistant Professor, Texas Woman's University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 19399
Record Dates: First submitted 2017-03-30; First posted 2017-04-25 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Masking Description: Investigator is blinded to intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Traction (Experimental): Intermittent lumbar traction will be performed in the prone position for 3 x 15-minute sessions at 40% of the participants body weight and will be adjusted based on the participants response.
  Interventions: Other: Lumbar traction

INTERVENTIONS:
Other: Lumbar traction — Lumbar traction is used to decompress the spinal structures and relieve pressure and may stretch the spine.

SUMMARY:
The objective in this study is to determine the predictive validity of a set of special clinical tests in identifying those who will respond to lumbar traction

DETAILED DESCRIPTION:
The objective in this study is to determine the predictive validity of a set of special clinical tests in identifying those who will respond to lumbar traction. The central hypothesis of this pilot study is that a cluster of lumbopelvic stress tests will be able to identify a subgroup of patients with low back pain who will respond favorably to mechanical lumbar traction. If these clinical tests can identify a subgroup of patients with low back pain who respond favorably to lumbar traction, additional studies, including randomized clinical trials will be necessary to further test and validate the use of this cluster of clinical tests. The rationale for this research is to examine the connection between provocative lumbar compression testing and lumbar traction as a means of decompression

ELIGIBILITY:
Inclusion Criteria:

* Complaints of low back pain with or without pain into the lower extremities
* Pain of at least 2/10 according to the Numeric Pain Rating Scale
* Score of at least 20 or greater on the Oswestry Disability Index

Exclusion Criteria:

* Medical red flags consistent with non-mechanical back pain (i.e. recent weight loss, history of cancer, night sweats, fever)
* Previous surgery to the lumbar spine
* Current pregnancy
* Any neurological symptoms in the lower extremities
* Evidence of central nervous system involvement
* The inability to lie prone for 15 minutes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-03-30 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Disability | 14 days
  Modified Oswestry Disability Index

SECONDARY OUTCOMES:
Change in Pain | 14 days
  Numeric Pain Rating Scale
Change in perceived outcome | 14 days
  Global Rating of Change

CONTACTS AND LOCATIONS:
Locations (1):
- Texas Woman's University-Dallas, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No